CLINICAL TRIAL: NCT03034954
Title: Effects of 3mA HD-tDCS on Associative and Working Memory in Cognitively Intact Older Adults
Brief Title: Patient Centered-Rehabilitation ver111090.1
Acronym: PCN1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Benjamin Hampstead, PhD, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00111090.1 PCN
Record Dates: First submitted 2016-10-24; First posted 2017-01-27 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Cognitive Change

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active HD-tDCS (Active Comparator): Participants will receive "real" HD-tDCS (3 milliamps for 20 minutes) for a single session.
  Interventions: Device: Active HD-tDCS
- Sham HD-tDCS (Sham Comparator): Participants will undergo the exact same procedures as the active group but will receive sham stimulation for a single session.
  Interventions: Device: Sham HD-tDCS

INTERVENTIONS:
Device: Active HD-tDCS — Participants will receive active HD-tDCS at 3mA for 20 minutes
  Other Names: HD-tDCS
  Arms: Active HD-tDCS
Device: Sham HD-tDCS — Participants will receive sham HD-tDCS
  Arms: Sham HD-tDCS

SUMMARY:
As we age, a number of factors can reduce our cognitive (or thinking) abilities. This study will evaluate whether transcranial electrical stimulation (TES), which uses small amounts of electricity to modulate brain functioning, can improve cognitive abilities. Here, the effects of TES on working memory, learning, and memory, will be evaluated in a group of healthy older adults.

DETAILED DESCRIPTION:
The primary objective is to investigate the cognitive effects of high definition anodal tDCS (HD-tDCS; anode at center electrode) at 3 mA (for 20 minutes) on learning, memory, and working memory. Participants will be randomized to active or sham stimulation and will complete a series of cognitive tests both during and after stimulation.

Tolerability and blinding will also be evaluated using standard side effect questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with intact cognitive functioning.
2. Participants will be age 50 or older.

Exclusion Criteria:

1. Individuals with a documented history of cognitive impairment.
2. A history of serious mental illness (e.g., bipolar disorder, schizophrenia, axis 2 disorders)
3. Sensory or motor impairments that limit the ability to take part in the study
4. A significant history or current use of alcohol or drug abuse/dependence
5. Those who are currently pregnant (if there is a question of pregnancy, pregnancy tests will be available for participants at no charge)
6. Participants with an Mini Mental State Examination score <24 at screening.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Hampstead, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan - Department of Psychiatry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were excluded after consent due to failing the tDCS safety screen. One participant endorsed a skin condition with lesions at site of electrode placement. One participant disclosed a prior head injury.
Period: Overall Study
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Started | 21 | 21
Completed | 20 | 21
Not Completed | 1 | 0
Not completed — Machine malfunction; did not reach 3 mA | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant was a statistical outlier for several behavioral measures and was excluded from baseline data and all analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Active HD-tDCS | Sham HD-tDCS | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.42 (8.546) | 65.38 (10.604) | 65.88 (9.573)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 21 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 40
Mini-Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — The Mini Mental-State Examination is a 30-item global cognitive screen. Scores range from 0-30 with higher scores represent better performances and scores 23 and below are suggestive of cognitive impairment. Population: Participants were not screened if an MMSE was completed within the past six months as part of their involvement with the Michigan Alzheimer's Disease Center (n = 2)
  units on a scale
    number analyzed (Participants) | 19 | 19 | 38
    (all) | 28.58 (1.216) | 28.37 (1.212) | 28.47 (1.202)
Education [Mean (Standard Deviation); unit: years] — Population: Missing data for two participants
  years
    number analyzed (Participants) | 17 | 21 | 38
    (all) | 16.82 (1.59) | 16.48 (2.089) | 16.63 (1.866)
Impedance [Mean (Standard Deviation); unit: quality units] — The first impedance reading averaged across all five electrodes. The unit measured is in "Quality Units" as produced by the Soterix transcranial direct current stimulation machine, which is a proprietary measurement of impedance. Lower values represent less impedance.
  quality units | 0.9512 (0.4004) | 0.8939 (.06314) | 0.921 (0.528)
Object Location Touchscreen Task (Version B) Free Recall Total Error [Mean (Standard Deviation); unit: centimeters] — The Object Location Touchscreen Task (OLTT) is an ecologically relevant measure of object location association memory. The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Free Recall, participants are given a black screen and asked to touch the area of the screen an object was located. Total Score is the sum of error for all 15 trials. Lower scores represent better performance.
  centimeters | 115.27 (44.445) | 102.534 (6.835) | 108.583 (7.239)
Object Location Touchscreen Task (Version B) Free Recall Average Error [Mean (Standard Deviation); unit: centimeters] — The Object Location Touchscreen Task (OLTT) is a measure of object location association memory. The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Free Recall, participants are given a blank screen and asked to touch the area of the screen an object was located. Average Score is the average error across all 15 trials. Lower scores represent better performance.
  centimeters | 7.685 (2.963) | 6.835 (2.97) | 7.239 (2.96)
Object Location Touchscreen Task (Version B) Free Recall Average Time to Respond [Mean (Standard Deviation); unit: milliseconds] — The Object Location Touchscreen Task (OLTT) is a measure of object location association memory. The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Free Recall, participants are given a blank screen and asked to touch the area of the screen an object was located. Average Time is the average latency to respond across all 15 trials. Lower scores represent faster responses.
  milliseconds | 3796.361 (1188.015) | 4921.558 (2306.631) | 4387.09 (1924.503)
Object Location Touchscreen Task (Version B) Cued Recall Total Error [Mean (Standard Deviation); unit: centimeters] — The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Cued Recall, participants are shown the "room" or environment on the screen and asked to touch the area of the screen an object was located. Total Score is the sum of error for all 15 trials. Lower scores represent better performance.
  centimeters | 74.513 (51.385) | 45.055 (38.61) | 59.048 (46.958)
Object Location Touchscreen Task (Version B) Cued Recall Average Error [Mean (Standard Deviation); unit: centimeters] — The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Cued Recall, participants are shown the "room" or environment on the screen and asked to touch the area of the screen an object was located. Average Score is the average error across all 15 trials. Lower scores represent better performance.
  centimeters | 4.971 (3.422) | 3.002 (2.574) | 3.937 (3.129)
Object Location Touchscreen Task (Version B) Cued Recall Average Time to Respond [Mean (Standard Deviation); unit: milliseconds] — The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Cued Recall, participants are shown the "room" or environment on the screen and asked to touch the area of the screen an object was located. Average Time is the average latency to respond across all 15 trials. Lower scores represent faster responses.
  milliseconds | 3855.83 (2452.1) | 3307.879 (1605.689) | 3568.155 (2043.063)
Object Location Touchscreen Task (Version B) Recognition Total Correct [Mean (Standard Deviation); unit: number of correct answers] — The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Recognition, participants are asked to select the correct location of an object from three options on the screen. Recognition total is the number of correct selections on all 15 trials. Higher scores represent better performance.
  number of correct answers | 13.11 (1.941) | 14.05 (1.322) | 13.6 (1.692)
Object Location Touchscreen Task (Version B) Recognition Average Time to Respond [Mean (Standard Deviation); unit: milliseconds] — The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Recognition, participants are asked to select the correct location of an object from three options on the screen. Recognition Average Response Time is the average latency to respond across all 15 trials. Lower scores represent faster responses.
  milliseconds | 3005.095 (1807.47) | 2456.063 (1164.46) | 2716.853 (1510.062)

OUTCOME MEASURES:

1. Primary Outcome: Object Location Touchscreen Task (Version C) Free Recall Total Error
Description: The Object Location Touchscreen Task (OLTT) is an ecologically relevant measure of object location association memory. The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Free Recall, participants are given a black screen and asked to touch the area of the screen an object was located. Total Score is the sum of error for all 15 trials. Lower scores represent better performance.
Time Frame: 15 minutes after encoding
Population: Missing data for one participant
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 20
centimeters | 121.498 (26.366) | 99.77 (27.845)
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; We used a multivariate statistic to compare OLTT means (Free Recall Total Error, Free Recall Average Error, Cued Recall Total Error, Cued Recall Average Error, Recognition Total Correct) at baseline (Version B) to post HD-tDCS OLTT means (Version C), by groups (active vs. sham). The overall statistic represents the simultaneous comparison of baseline OLTT measures to post HD-tDCS OLTT measures; Test type: Other; p = .300, Repeated Measures ANOVA — Reported p-value represents Time (baseline to post-tDCS) x Condition (Active or Sham) interaction for all OLTT Accuracy Measures. If the multivariate statistic is not significant no univariate statistical analyses are completed; repeated measures (OLTT baseline and post-tDCS); between-subjects (active vs. sham)

2. Primary Outcome: Object Location Touchscreen Task (Version C) Free Recall Average Error
Description: The Object Location Touchscreen Task (OLTT) is a measure of object location association memory. The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Free Recall, participants are given a blank screen and asked to touch the area of the screen an object was located. Average Score is the average error across all 15 trials. Lower scores represent better performance.
Time Frame: 15 minutes after encoding
Population: Missing data for one participant
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 20
centimeters | 8.099 (1.757) | 6.652 (1.856)

3. Primary Outcome: Object Location Touchscreen Task (Version C) Free Recall Average Time to Respond
Description: The Object Location Touchscreen Task (OLTT) is a measure of object location association memory. The OLTT requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Free Recall, participants are given a blank screen and asked to touch the area of the screen an object was located. Average Time is the average latency to respond across all 15 trials. Lower scores represent faster responses.
Time Frame: 15 minutes after encoding
Population: Missing data for one participant
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 20
milliseconds | 3419.878 (1690.354) | 3029.648 (1572.416)
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; A Repeated Measures ANOVA was used to compare baseline OLTT (Version B) to post-tDCS OLTT (Version C) across the treatment groups (Active vs. Sham). The multivariate analyses included OLTT Response Times (i.e., Free Recall Average Response Time, Cued Recall Average Response Time, Recognition Average Response Time); Test type: Other; p = .044, Repeated Measures ANOVA — Statistic represents the interaction between Time (baseline to post-tDCS) by Condition (Active vs. Sham)
Statistical Analysis 2: Comparison: Active HD-tDCS vs Sham HD-tDCS; Univariate analysis of the OLTT Free Recall Average Time to Respond following significant multivariate repeated measures ANOVA comparing baseline OLTT (Version B) to post-tDCS OLTT (Version C) across the treatment groups (Active vs. Sham); Test type: Other; p = .006, Repeated Measures ANOVA

4. Primary Outcome: Object Location Touchscreen Task (Version C) Cued Recall Total Error
Description: The Object Location Touchscreen Task (OLTT) requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Cued Recall, participants are shown the "room" or environment on the screen and asked to touch the area of the screen an object was located. Total Score is the sum of error for all 15 trials. Lower scores represent better performance.
Time Frame: 15 minutes after encoding
Population: Missing data for one participant
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 20
centimeters | 66.806 (29.303) | 43.775 (29.32)

5. Primary Outcome: Object Location Touchscreen Task (Version C) Cued Recall Average Error
Description: The Object Location Touchscreen Task (OLTT) requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Cued Recall, participants are shown the "room" or environment on the screen and asked to touch the area of the screen an object was located. Average Score is the average error across all 15 trials. Lower scores represent better performance.
Time Frame: 15 minutes after encoding
Population: Missing data for one participant
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 20
centimeters | 4.453 (1.954) | 2.919 (1.954)

6. Primary Outcome: Object Location Touchscreen Task (Version C) Cued Recall Average Time to Respond
Description: The Object Location Touchscreen Task (OLTT) requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Cued Recall, participants are shown the "room" or environment on the screen and asked to touch the area of the screen an object was located. Average Time is the average latency to respond across all 15 trials. Lower scores represent faster responses.
Time Frame: 15 minutes after encoding
Population: Missing data for one participant
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 20
milliseconds | 3991.659 (2218.596) | 2666.858 (866.887)
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Univariate analysis of the OLTT Cued Recall Average Time to Respond following significant multivariate repeated measures ANOVA comparing baseline OLTT (Version B) to post-tDCS OLTT (Version C) across the treatment groups (Active vs. Sham); Test type: Other; p = .15, Repeated Measures ANOVA

7. Primary Outcome: Object Location Touchscreen Task (Version C) Recognition Total Correct
Description: The Object Location Touchscreen Task (OLTT) requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Recognition, participants are asked to select the correct location of an object from three options on the screen. Recognition total is the number of correct selections on all 15 trials. Higher scores represent better performance.
Time Frame: 15 minutes after encoding
Population: Missing data for one participant
Measure: Mean (Standard Deviation); unit: number of correct answers
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 20
number of correct answers | 12.79 (1.932) | 13.45 (1.669)

8. Primary Outcome: Object Location Touchscreen Task (Version C) Recognition Average Time to Respond
Description: The Object Location Touchscreen Task (OLTT) requires participants to learn and recall the location of 15 object-location associations. Memory is evaluated using a touchscreen monitor, which allows for the continuous measurement of memory accuracy (i.e., distance from targeted location). During the Recognition, participants are asked to select the correct location of an object from three options on the screen. Recognition Average Response Time is the average latency to respond across all 15 trials. Lower scores represent faster responses.
Time Frame: 15 minutes after encoding
Population: Missing data for one participant
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 20
milliseconds | 2804.459 (1244.249) | 1903.39 (843.244)
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Univariate analysis of the OLTT Recognition Average Time to Respond following significant multivariate repeated measures ANOVA comparing baseline OLTT (Version B) to post-tDCS OLTT (Version C) across the treatment groups (Active vs. Sham); Test type: Other; p = .3, Repeated Measures ANOVA

9. Primary Outcome: Performance (d') on a Simple Attention (0-back) Test
Description: The n-back is a well validated measure of working memory. During 0-back, participants are asked to respond by pressing a key when the picture on the screen is the same as the given target (e.g., a cow). Discriminability (d') is a measure of signal detection that accounts for signal to noise ratio. Higher scores represent better discriminability.
Time Frame: 30 minutes post-stimulation
Population: missing data for two participants
Measure: Mean (Standard Deviation); unit: d'
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 17 | 21
d' | 4.26 (.231) | 4.25 (.219)

10. Primary Outcome: Performance (d') on a Working Memory (2-back) Test
Description: The n-back is a well validated measure of working memory. During 2-back, participants are asked to respond when a picture shown is the exact same as two items ago. Discriminability (d') is a measure of signal detection that accounts for signal to noise ratio. Higher scores represent better discriminability.
Time Frame: 30 minutes post-stimulation
Population: missing data for two participants
Measure: Mean (Standard Deviation); unit: d'
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 17 | 21
d' | 3.05 (.508) | 2.94 (.675)

11. Primary Outcome: Performance (d') on a Working Memory (Semantic 2-back) Test
Description: The n-back is a well validated measure of working memory. During Semantic-back, participants are asked to respond when a picture shown is in the same semantic category as the picture two items ago (e.g., both fruits). Discriminability (d') is a measure of signal detection that accounts for signal to noise ratio. Higher scores represent better discriminability.
Time Frame: 30 minutes post-stimulation
Population: missing data for eleven participants (5 Active; 6 Sham) due to Eprime miscalculation
Measure: Mean (Standard Deviation); unit: d'
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 14 | 15
d' | 1.518 (.537) | 1.69 (.495)

12. Primary Outcome: Calculated Working Memory Performance Accounting for Simple Attention (2-back d' Minus 0-back d')
Description: The n-back is a well validated measure of working memory. During 0-back, participants are asked to respond by pressing a key when the picture on the screen is the same as the given target (e.g., a cow). During 2-back, participants are asked to respond when a picture shown is the exact same as two items ago. Discriminability (d') is a measure of signal detection that accounts for signal to noise ratio. By subtracting the 0-back d', the calculated score represents a more pure working memory measure. Scores closer to zero or positive represent better working memory performance.
Time Frame: 30 minutes post-stimulation
Population: missing data for 12 participants: 11 2-back (5 Active; 6 sham) due to Eprime miscalculation & one 0-back (Active)
Measure: Mean (Standard Deviation); unit: d'
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 13 | 15
d' | -1.130 (.629) | -1.31 (.675)

13. Primary Outcome: Calculated Working Memory Performance Accounting for Simple Attention (Semantic 2-back d' Minus 0-back d')
Description: The n-back is a well validated measure of working memory. During 0-back, participants are asked to respond by pressing a key when the picture on the screen is the same as the given target (e.g., a cow). During Semantic 2-back, participants are asked to respond when a picture shown is in the same semantic category as the picture two items ago (e.g., both fruits). Discriminability (d') is a measure of signal detection that accounts for signal to noise ratio. By subtracting the 0-back d', the calculated score represents a more pure working memory measure. Scores closer to zero or positive represent better working memory performance.
Time Frame: 30 minutes post-stimulation
Population: missing data for two participants
Measure: Mean (Standard Deviation); unit: d'
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 17 | 21
d' | -2.69 (.58) | -2.56 (.47)
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; A Multivariate ANOVA was used to compare Active vs. Sham groups on discriminability measures (i.e. 0-back d', 2-back d', semantic 2-back d') and calculated working memory measures (i.e., 2-back d' minus 0-back d', semantic 2-back d' minus 0-back d'); Test type: Other; p = .450, MANOVA

14. Secondary Outcome: Blinding in Total Sample
Description: Participants were asked to estimate which group they were in (i.e., active or sham).
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  Said Active | 9 | 6
  Said Sham | 9 | 8
  Said Don't Know | 1 | 7
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Chi-squared tests were conducted to determine group differences in actual condition assignment vs. estimated/perceived condition; Test type: Other; p = .078, Chi-squared

15. Secondary Outcome: Frequency of Endorsement (%) for Headache Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: The side effects were assessed using a modified version of Brunoni et al. (2011) questionnaire. Participants rated common sensory experiences on a scale of "None, Mild, Moderate, or Severe".
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  Headache NONE | 19 | 18
  Headache MILD | 0 | 3
  Headache MODERATE | 0 | 0
  Headache SEVERE | 0 | 0
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Test type: Other; p = .233, Fisher Exact

16. Secondary Outcome: Frequency of Endorsement (%) for Neck Pain Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: as for outcome 15
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  Neck Pain NONE | 19 | 21
  Neck Pain MILD | 0 | 0
  Neck Pain MODERATE | 0 | 0
  Neck Pain SEVERE | 0 | 0

17. Secondary Outcome: Frequency of Endorsement (%) for Scalp Pain Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: as for outcome 15
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  NONE | 16 | 20
  MILD | 1 | 0
  MODERATE | 1 | 1
  SEVERE | 1 | 0
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Test type: Other; p = .600, Fisher Exact

18. Secondary Outcome: Frequency of Endorsement (%) for Tingling Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: as for outcome 15
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  NONE | 6 | 7
  MILD | 12 | 11
  MODERATE | 1 | 2
  SEVERE | 0 | 1
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Test type: Other; p = .999, Fisher Exact

19. Secondary Outcome: Frequency of Endorsement (%) for Itching Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: as for outcome 15
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  NONE | 16 | 14
  MILD | 3 | 7
  MODERATE | 0 | 0
  SEVERE | 0 | 0
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Test type: Other; p = .281, Fisher Exact

20. Secondary Outcome: Frequency of Endorsement (%) for Burning Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: as for outcome 15
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  NONE | 9 | 7
  MILD | 10 | 8
  MODERATE | 0 | 5
  SEVERE | 0 | 1
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Test type: Other; p = .082, Fisher Exact

21. Secondary Outcome: Frequency of Endorsement (%) for Skin Redness Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: as for outcome 15
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  NONE | 19 | 19
  MILD | 0 | 2
  MODERATE | 0 | 0
  SEVERE | 0 | 0
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Test type: Other; p = .490, Fisher Exact

22. Secondary Outcome: Frequency of Endorsement (%) for Sleepiness Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: as for outcome 15
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  NONE | 19 | 18
  MILD | 0 | 2
  MODERATE | 0 | 1
  SEVERE | 0 | 0
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Test type: Other; p = .488, Fisher Exact

23. Secondary Outcome: Frequency of Endorsement (%) for Concentration Changes Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: as for outcome 15
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  NONE | 17 | 21
  MILD | 2 | 0
  MODERATE | 0 | 0
  SEVERE | 0 | 0
Statistical Analysis 1: Comparison: Active HD-tDCS vs Sham HD-tDCS; Test type: Other; p = .219, Fisher Exact

24. Secondary Outcome: Frequency of Endorsement (%) for Mood Changes Item in Active and Sham Participants Undergoing HD-tDCS Session
Description: as for outcome 15
Time Frame: ~1 minute post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 19 | 21
Participants
  NONE | 19 | 21
  MILD | 0 | 0
  MODERATE | 0 | 0
  SEVERE | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for the duration of participation (i.e., approximately 2-3 hours)
Arm/Group | Active HD-tDCS | Sham HD-tDCS
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 16/19 | 19/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active HD-tDCS (N=19) | Sham HD-tDCS (N=21)
Headache (General disorders) | 0 (0) | 3 (3)
Neck Pain (General disorders) | 0 (0) | 0 (0)
Scalp Pain (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Tingling (Skin and subcutaneous tissue disorders) | 13 (13) | 14 (14)
Itching (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7)
Burning sensation (Skin and subcutaneous tissue disorders) | 10 (10) | 14 (14)
Skin redness (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Sleepiness (General disorders) | 0 (0) | 3 (3)
Concentration Changes (General disorders) | 2 (2) | 0 (0)
Mood Changes (Psychiatric disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT03034954/Prot_SAP_000.pdf